CLINICAL TRIAL: NCT06890728
Title: SPICE UP MyPlate - Strategy for Promoting Intake of Delicious Healthful Dietary Patterns Based on MyPlate: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Kristina Petersen PhD, APD, FAHA, Associate Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SUP
Record Dates: First submitted 2025-03-17; First posted 2025-03-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Cardiometabolic Risk Factors
Keywords: diet quality; nutrition education; culinary medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culinary focused nutrition education (Experimental): The intervention group will receive a 12-week culinary focused nutrition education program. Participants in the intervention group will receive culinary focused nutrition education based on MyPlate with an emphasis on taste and enjoyment of healthy foods. Using herbs and spices to flavor foods will be the emphasis. The intervention will be delivered in an online format with online content delivery . The intervention will consist of eight modules. Modules one to four will be provided during the first month. Modules four to eight will be provided during months 2 and 3.
  Interventions: Behavioral: Culinary focused nutrition education
- Standard nutrition education (Active Comparator): The control group will represent standard low intensity nutrition education. Control group participants will be provided with a printed MyPlate resource.
  Interventions: Behavioral: Standard low intensity nutrition education

INTERVENTIONS:
Behavioral: Culinary focused nutrition education — Culinary focused nutrition education based on MyPlate with an emphasis on taste and enjoyment of healthy foods.
  Arms: Culinary focused nutrition education
Behavioral: Standard low intensity nutrition education — Provided by a written MyPlate resource
  Arms: Standard nutrition education

SUMMARY:
The aim is to conduct a pilot study to assess the feasibility, acceptability and potential effectiveness of culinary focused nutrition education to promote increased adherence to the Dietary Guidelines for Americans compared to standard low-intensity care.

DETAILED DESCRIPTION:
This is a 15-week, 2-arm randomized controlled pilot trial. In a 1:1 ratio, participants will be randomized to the intervention arm or the control arm. The intervention group will receive a 12-week culinary focused nutrition education program. The control group will receive standard low-intensity care (i.e., printed healthy eating material). Outcome measures will be assessed at baseline and 15 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 31-59 years
* Involved in meal cooking at home and consumes a home cooked meal ≥ 1 time per week
* Individuals taking medications for blood pressure, lipid or glucose lowering will be eligible if they have been on a stable dose for the 1 month prior to baseline

Exclusion Criteria:

* A member of the household is already enrolled (only one person per household will be eligible for inclusion in the study).
* Unstable medical conditions requiring active intervention (surgeries, medication/drug therapy for < 3 months) as assessed during the telephone screening (e.g. cancer, kidney disease requiring dialysis, heart or gastrointestinal diseases requiring surgery).
* Received nutrition education for a medical condition within the past 6 months
* Currently following a weight loss diet
* Lost ≥ 10% body weight in the past 6 months
* Currently (within 6 months) smoke or use any tobacco or nicotine containing products
* Currently pregnant or given birth within the prior 6 months
* Currently participating in another clinical trial
* Principal investigator discretion (e.g., disrespectful or inappropriate interactions with study staff)
* Does not speak or understand English

Ages: 31 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Diet quality change | 15 weeks
  Change in diet quality assessed by the Healthy Eating Index-2015 (HEI-2015) assessed by 24-hour recalls

SECONDARY OUTCOMES:
Diet quality component scores change | 15 weeks
  Change in the 13 components that comprise the Healthy Eating Index-2015 (HEI-2015) assessed by 24 hour recalls
Food group intake change | 15 weeks
  Changes in intake of fruits; vegetables; refined grains; wholegrains; dairy; meat, poultry, eggs; seafood; nuts, seeds and soy products; oils) assessed by 24-hour recalls
Change in intake of added sugars, sodium and saturated fat | 15 weeks
  Changes in intake of added sugars, sodium and saturated fat assessed by 24 hour recalls
Change in weight | 15 weeks
  assessed by electronic scale
Change in waist circumference | 15 weeks
  Assessed by tape measure at 1 cm above the naval
Change in central systolic and diastolic blood pressure | 15 weeks
  Assessed using a SphymoCor Xcel (Atcor Medical)
Change in brachial systolic and diastolic blood pressure | 15 weeks
  Blood pressure measured assessed using a SphymoCor Xcel (Atcor Medical)
Change in carotid-femoral pulse wave velocity | 15 weeks
  Assessed using a SphymoCor Xcel (Atcor Medical)
Change in LDL-cholesterol | 15 weeks
  Assessed from fasting blood draw expressed in mg/dL. LDL-cholesterol will be measured directly via enzymatic assay.
Change in total cholesterol | 15 weeks
  Assessed from fasting blood draw expressed in mg/dL.
Change in HDL-Cholesterol | 15 weeks
  Assessed from fasting blood draw expressed in mg/dL.
Change in triglycerides | 15 weeks
  Assessed from fasting blood draw expressed in mg/dL.
Change in fasting glucose | 15 weeks
  Assessed in a fasting blood draw and expressed in mg/dL
Change in HbA1c | 15 weeks
  Assessed in a fasting blood draw and expressed in %
Program acceptability and satisfaction | 15 weeks
  Assessed via surveys

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Petersen, PhD, Principal Investigator — Penn State University
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP
Time Frame: Statistical analysis plan will be uploaded before database lock and unblinding of randomization codes

DOCUMENTS (1):
  • Statistical Analysis Plan (2026-01-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT06890728/SAP_000.pdf